CLINICAL TRIAL: NCT00614445
Title: A Double-Blind, Multicenter, Randomized, Placebo-Controlled Trial Of The Efficacy Of Diclectin® For Nausea And Vomiting Of Pregnancy
Brief Title: The Efficacy Of Diclectin® For Nausea And Vomiting Of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duchesnay Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIC-301
Record Dates: First submitted 2008-01-29; First posted 2008-02-13 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2011-08

CONDITIONS: Nausea and Vomiting of Pregnancy
Keywords: Nausea; Vomiting; Pregnancy; Hyperemesis gravidarum; Pregnancy complications
MeSH Terms: conditions — Nausea; Vomiting; Hyperemesis Gravidarum; Pregnancy Complications | interventions — doxylamine succinate; Pyridoxine; dicyclomine, doxylamine, pyridoxine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclectin® (Experimental): Diclectin® (doxylamine succinate 10 mg and pyridoxine hydrochloride 10 mg) delayed release tablet
  Interventions: Drug: doxylamine succinate 10 mg/pyridoxine hydrochloride 10 mg
- Placebo (Placebo Comparator): Placebo tablets identical in size, shape, taste, and color to the experimental treatment (Diclectin®)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: doxylamine succinate 10 mg/pyridoxine hydrochloride 10 mg — up to 4 tablets daily, titrated according to the protocol
  Other Names: Diclectin®
  Arms: Diclectin®
Drug: Placebo — 2 to 4 tablets daily titrated according to the protocol
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Diclectin® (doxylamine succinate USP 10 mg and pyridoxine HCl 10 mg) is more effective at controlling the nausea and vomiting of pregnancy than a placebo.

DETAILED DESCRIPTION:
Nausea and vomiting of pregnancy (NVP), also known as "morning sickness," is a common condition that affects a large percentage of pregnant women. The symptoms can range from mild nausea to severe nausea and vomiting for which a woman may need to be hospitalized. Nausea and vomiting of pregnancy can affect a woman's quality of life and ability to conduct daily activities.

Diclectin® is a combination of 10 mg doxylamine succinate (an antihistamine), and 10 mg pyridoxine hydrochloride (vitamin B6) in a delayed release tablet formulation. It has been commercially available in Canada for the management of NVP for over 25 years and has been prescribed to over 33 million pregnant women.

Presently, there is no Food Drug and Administration (FDA) approved drug on the market to treat the symptoms of NVP. This study will test the efficacy of Diclectin® (doxylamine 10 mg, pyridoxine 10 mg in a delayed-release formulation) for NVP.

Patients enrolled in the study will receive between 2 and 4 tablets of Diclectin® or placebo daily, depending on their symptoms for up to 14 days. Patients will assess their symptoms of nausea and vomiting daily using a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed a written informed consent to participate in the study and has agreed to follow dosing instructions and complete all required study visits.
* The patient is a pregnant female age equal to or greater than 18 years old.
* The patient's entry ultrasound indicates a viable pregnancy and confirms gestational age of the fetus is 7-14 weeks at the anticipated time of the first dose of study medication or placebo. If an ultrasound was done within 4 weeks of the admission visit, and results can be obtained, an additional ultrasound is not necessary.
* The patient is suffering from NVP and has a Pregnancy Unique Quantification of Emesis (PUQE) score ≥6.
* The patient has not responded to conservative management consisting of dietary/lifestyle advice according to the 2004 ACOG Practice Bulletin.
* The patient agrees, if on a multivitamin, to continue on their current dose of multivitamin for the duration of the trial.
* The patient does not plan termination of the pregnancy.

Exclusion Criteria:

* The investigator confirms the patient's nausea and vomiting is of etiology other than Nausea and Vomiting of Pregnancy (NVP).
* The patient has gestational trophoblastic disease or multifetal gestation.
* The patient has a condition for which antihistamines, in the opinion of the investigator, are contraindicated (epilepsy, alcoholism, glaucoma, chronic lung disease, urinary retention, heart block, etc.).
* The patient has used antihistamines, anticholinergics, dopamine antagonists, serotonin antagonists, ginger, or anti-emetic therapy (including acupressure, acupuncture, homeopathic remedies, medical hypnosis, relief bands etc) to treat NVP in the previous 48 hours or plans to do so during the study .
* The patient is using drugs that have anticholinergic activity (e.g., tricyclic antidepressants).
* The patient is taking multivitamins containing more than 10 mg of vitamin B6, or plans to do so during the study.
* The patient is taking supplementary vitamin B6 in addition to any multivitamin preparation, or plans to do so during the study.
* The patient is currently drinking any amount of alcohol.
* The patient has any condition that might interfere with the conduct of the study.
* The patient is likely to be unable to comply with study procedures because of inadequate cognitive skills.
* The patient has received an investigational drug within 30 days before enrollment in this study or is scheduled to receive an investigational drug during the course of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liubov Gargaun, M.D., Study Director — Duchesnay Inc.; Gideon Koren, M.D., Principal Investigator — Motherisk Program, University of Toronto; Gary Hankins, M.D., Principal Investigator — University of Texas
Locations (7):
- United States (7):
  - Washington Hospital Center Physicians, Washington D.C., District of Columbia
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - National Naval Medical Center, Bethesda, Maryland
  - Magee-Womens Hospital of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Pasadena Clinic, Pasadena, Texas
  - UTMB Regional Maternal & Child Health Program--Pearland Clinic, Pearland, Texas

REFERENCES:
- [Derived] Persaud N, Meaney C, El-Emam K, Moineddin R, Thorpe K. Doxylamine-pyridoxine for nausea and vomiting of pregnancy randomized placebo controlled trial: Prespecified analyses and reanalysis. PLoS One. 2018 Jan 17;13(1):e0189978. doi: 10.1371/journal.pone.0189978. eCollection 2018. PMID 29342163
- [Derived] Koren G, Clark S, Hankins GD, Caritis SN, Umans JG, Miodovnik M, Mattison DR, Matok I. Demonstration of early efficacy results of the delayed-release combination of doxylamine-pyridoxine for the treatment of nausea and vomiting of pregnancy. BMC Pregnancy Childbirth. 2016 Nov 24;16(1):371. doi: 10.1186/s12884-016-1172-9. PMID 27881103
- [Derived] Koren G, Hankins GD, Clark S, Caritis SN, Miodovnik M, Umans JG, Mattison DR. Effectiveness of doxylamine-pyridoxine for morning sickness. Am J Obstet Gynecol. 2016 May;214(5):664-6. doi: 10.1016/j.ajog.2016.01.186. Epub 2016 Feb 1. No abstract available. PMID 26844757
- [Derived] Koren G, Clark S, Hankins GD, Caritis SN, Umans JG, Miodovnik M, Mattison DR, Matok I. Maternal safety of the delayed-release doxylamine and pyridoxine combination for nausea and vomiting of pregnancy; a randomized placebo controlled trial. BMC Pregnancy Childbirth. 2015 Mar 18;15:59. doi: 10.1186/s12884-015-0488-1. PMID 25884778
- [Derived] Matok I, Clark S, Caritis S, Miodovnik M, Umans JG, Hankins G, Mattison DR, Koren G. Studying the antiemetic effect of vitamin B6 for morning sickness: pyridoxine and pyridoxal are prodrugs. J Clin Pharmacol. 2014 Dec;54(12):1429-33. doi: 10.1002/jcph.369. Epub 2014 Aug 7. PMID 25052410
- [Derived] Costantine MM, Matok I, Chiossi G, Clark S, Miodovnik M, Umans JG, Caritis S, Hankins GD, Koren G. Determinants of adherence to delayed-release doxylamine and pyridoxine in patients with nausea and vomiting of pregnancy. Ther Drug Monit. 2012 Oct;34(5):569-73. doi: 10.1097/FTD.0b013e31826e7997. PMID 22972538
- [Derived] Koren G, Clark S, Hankins GD, Caritis SN, Miodovnik M, Umans JG, Mattison DR. Effectiveness of delayed-release doxylamine and pyridoxine for nausea and vomiting of pregnancy: a randomized placebo controlled trial. Am J Obstet Gynecol. 2010 Dec;203(6):571.e1-7. doi: 10.1016/j.ajog.2010.07.030. Epub 2010 Sep 16. PMID 20843504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a double-blind, randomized, multicenter, placebo-controlled study in the treatment of NVP. On Day 1, all patients will receive 2 tablets of study drug at bedtime. During Days 2-14 the patients will receive 2 tablets of study drug at bedtime plus additional study drug based upon the need for control of their nausea and vomiting.
Pre-assignment Details: The minimum dosage will be 2 tablets daily at bedtime, increasing, when indicated, to the maximal dosage of 4 tablets per day. After randomization, patients will return to the clinic for evaluation on Day 4 (+/-1 day) and Day 8 (+/-1 day), and will return on Day 15 (+/-1 day) for an end of study visit. The study duration is expected to be 15 days.
Period: Overall Study
Arm/Group | Diclectin® | Placebo
Started | 140 | 140
Completed | 112 | 91
Not Completed | 28 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclectin® | Placebo | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 140 | 140 | 280
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (6.0) | 25.0 (5.6) | 25.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 140 | 280
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 140 | 140 | 280

OUTCOME MEASURES:

1. Primary Outcome: Diclectin Versus Placebo for Treatment of Nausea and Vomiting of Pregnancy (NVP) as Measured by the Change in Pregnancy Unique-Quantification of Emesis (PUQE) Overall Score of Symptoms From Baseline (Day 1) to End of Study Visit (Day 15).
Description: The objective of this double-blind, randomized, placebo-controlled study was to assess the efficacy, safety, and tolerability of oral Diclectin® in the treatment of nausea and vomiting of pregnancy (NVP) as measured by the Pregnancy Unique-Quantification of Emesis (PUQE) overall score of symptoms from baseline (Day 1) to end of study visit (Day 15). The PUQE score measured hours of nausea, number of times vomiting, and number of times retching for a TOTAL overall score of symptoms on a scale rated from 3 (no symptoms) to 15 (most severe).
Time Frame: Baseline (Day 1) to End of Study Visit Day 15 (± 1 day)
Population: Planned: Approximately 280 subjects (140 subjects per treatment group) were to be enrolled to achieve 200 evaluable subjects. Analyzed: 280 enrolled subjects [261 subjects in the intent-to-treat safety (ITT-S) population; 256 subjects in the intent-to-treat efficacy (ITT-E) population].
Measure: Mean (95% Confidence Interval); unit: PUQE Score
Arm/Group | Diclectin® | Placebo
Number analyzed (Participants) | 140 | 140
PUQE Score | -4.8 [-5.26 to -4.34] | -3.9 [-4.36 to -3.44]

ADVERSE EVENTS:
Arm/Group | Diclectin® | Placebo
Serious Adverse Events (participants affected / at risk) | 4/133 | 5/128
Other Adverse Events (participants affected / at risk) | 65/133 | 63/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclectin® (N=133) | Placebo (N=128)
Intra-uterine Death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Premature rupture of membrane (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Foetal disorder (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclectin® (N=133) | Placebo (N=128)
Adominal Pain (Gastrointestinal disorders) | 5 (5) | 8 (8)
Fatigue (General disorders) | 9 (9) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Dizziness (Nervous system disorders) | 8 (8) | 8 (8)
Headache (Nervous system disorders) | 17 (17) | 20 (20)
Somnolence (Nervous system disorders) | 19 (19) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished data given to the investigator may be transmitted to a third party without prior approval of the sponsor in writing. No publications or communications involving the results of the trial are authorized without prior review and written consent from the sponsor. The investigator must agree to send the sponsor for review prior to their submission. The sponsor reserves the right to delete from such materials any part or parts deemed to be confidential or proprietary.